CLINICAL TRIAL: NCT05961371
Title: Strength Training for Osteoporosis Prevention During Early Menopause
Acronym: STOP-EM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Leigh Gabel, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB22-1632
Record Dates: First submitted 2023-06-26; First posted 2023-07-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Bone Loss; Bone Loss, Age-related; Osteoporosis; Musculoskeletal Diseases
Keywords: Exercise; Resistance Training; Strength Training
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Musculoskeletal Diseases; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to the exercise or waitlist control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors will be masked to the group allocation of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): In-person, supervised resistance training program
  Interventions: Other: Resistance Training
- Control (No Intervention): Waitlist control group. Will be offered the exercise program following a 9-month wait.

INTERVENTIONS:
Other: Resistance Training — Twice weekly resistance training progressing to 5 sets of 5 repetitions of 80-90% of one repetition maximum.
  Arms: Exercise

SUMMARY:
The goal of this clinical pilot trial is to learn about the feasibility of a high-intensity resistance training intervention in peri- and early menopausal females. The main question it aims to answer are:

-Is a 9-month resistance training intervention feasible (e.g., recruitment rates, protocol adherence, attrition)

Secondary aims include examining changes in bone health, muscle strength, and menopausal symptoms.

Participants will participate in a 9-month progressive, supervised, resistance training intervention. Researchers will compare secondary outcomes between the exercise group and a wait-list control group.

DETAILED DESCRIPTION:
The STOP-EM trial will examine a 9-month supervised, progressive, resistance training program in peri- and early menopausal females. Primary outcomes include recruitment rates, protocol adherence, and attrition. A waitlist control group will allow us to examine the effect of the exercise program on bone density, structure, and strength, muscle strength, and menopausal symptoms. Participants will be randomized to the exercise or control group. The exercise group will attend twice weekly, in-person, supervised, progressive resistance training and build up to 80-90% of estimated 1 repetition maximum (1RM). The study will take place at the University of Calgary. Findings will be used to decide whether to continue to the definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* 45-60 years old.
* Menopause status of peri- or early menopausal: stages -2 or -1 of the stages for reproductive aging 10+ staging system or are within 5 years of their last known menses.

Exclusion Criteria:

* Females who are pregnant or planning pregnancy within the next year.
* Orthopaedic conditions that may be made worse with exercise.
* Has low back pain, hypertension, lipidemia, diabetes, or cardiovascular disease.
* Has a history of metabolic bone disease.
* Has had an osteoporotic fracture within the last 5 years.
* Had previous treatment with osteoporosis pharmacotherapy.
* Has active glucocorticoid use.
* Is currently participating in progressive resistance training or has in the previous 6 months.
* Has low serum vitamin D (25(OH)D) < 30 nmol/L or serum calcium <2.10 mmol/L.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | Over 9 months
  Recruitment rates - number of participants recruited per month and number of eligible participants who consented.
Feasibility - Adherence | Over 9 months
  Protocol adherence (number of exercise sessions participants attend) will be expressed as a percent.
Feasibility - Attrition | Over 9 months
  Attrition (number of randomized participants with valid outcome data) will be expressed as a percent.

SECONDARY OUTCOMES:
Volumetric bone mineral density (BMD) | Baseline and 9 months
  High-resolution peripheral quantitative computed tomography (HR-pQCT) will assess total, trabecular, and cortical BMD in mg/cm^3 at the distal tibia and radius.
Bone microarchitecture | Baseline and 9 months
  HR-pQCT will assess trabecular thickness and separation and cortical bone thickness in mm at the distal tibia and radius.
Bone strength | Baseline and 9 months
  Finite element analysis will be applied to HR-pQCT images at the distal tibia and radius to estimate bone strength (failure load) in N.
areal bone mineral density | Baseline and 9 months
  Dual X-ray absorptiometry (DXA) will measure areal bone mineral density (aBMD) in mg/cm^2 for the left hip (total hip and femoral neck), lumbar spine, and whole body.
Muscle strength | Baseline and 9 months
  Muscle strength testing will include max voluntary contractions of the knee extensors using an isometric dynamometer. Hand grip strength will be measured using a handgrip dynamometer.
Balance | Baseline and 9 months
  The four-square-step test assesses dynamic balance.
Aerobic Fitness | Baseline and 9 months
  The 6-minute walk test assesses aerobic fitness
Estrogen concentration | Baseline and 9 months
  A blood sample will measure plasma estradiol in pmol/L
Follicle stimulating hormone concentration | Baseline and 9 months
  A blood sample will measure plasma follicle stimulating hormone (FSH) in IU/L
Vitamin D concentration | Baseline and 9 months
  A blood sample will measure plasma 25-hydroxyvitamin D in nmol/L
Calcium concentration | Baseline and 9 months
  A blood sample will measure plasma calcium in mmol/L
Creatinine concentration | Baseline and 9 months
  A blood sample will measure plasma creatinine in umol/L
Biomarker of bone resorption | Baseline and 9 months
  A blood sample will measure plasma c-telopeptide (CTx) in ng/L
Biomarker of bone formation | Baseline and 9 months
  A blood sample will measure plasma procollagen 1 intact N-terminal propeptide (P1NP) in ug/L
Physical activity | Baseline and 9 months
  Physical activity will be assessed by wearing an accelerometer for 7 days to assess moderate to vigorous physical activity in minutes per day.
Menopausal quality of life | Baseline and 9 months
  Menopausal symptoms will be evaluated through the menopause-specific quality of life questionnaire with a minimum score of 0 and maximum score of 174 and a higher score indicating poorer outcomes
Menopausal symptoms | 9 months
  Menopausal symptoms will be evaluated through the menopause symptoms treatment satisfaction questionnaire with a minimum score of 0 and maximum score of 40 and a higher score indicating poorer outcomes
Body mass | Baseline and 9 months
  Body mass in kg
Height | Baseline and 9 months
  Height in cm

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Gabel, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson S, Weeks B, Weis L, Harding A, Horan S, Beck B. High-Intensity Resistance and Impact Training Improves Bone Mineral Density and Physical Function in Postmenopausal Women With Osteopenia and Osteoporosis: The LIFTMOR Randomized Controlled Trial. J Bone Miner Res. 2019 Mar;34(3):572. doi: 10.1002/jbmr.3659. Epub 2019 Feb 25. No abstract available. PMID 30861219
- [Background] Kistler-Fischbacher M, Weeks BK, Beck BR. The effect of exercise intensity on bone in postmenopausal women (part 2): A meta-analysis. Bone. 2021 Feb;143:115697. doi: 10.1016/j.bone.2020.115697. Epub 2020 Dec 24. PMID 33357834
- [Background] Lewis M, Bromley K, Sutton CJ, McCray G, Myers HL, Lancaster GA. Determining sample size for progression criteria for pragmatic pilot RCTs: the hypothesis test strikes back! Pilot Feasibility Stud. 2021 Feb 3;7(1):40. doi: 10.1186/s40814-021-00770-x. PMID 33536076
- [Background] Finkelstein JS, Brockwell SE, Mehta V, Greendale GA, Sowers MR, Ettinger B, Lo JC, Johnston JM, Cauley JA, Danielson ME, Neer RM. Bone mineral density changes during the menopause transition in a multiethnic cohort of women. J Clin Endocrinol Metab. 2008 Mar;93(3):861-8. doi: 10.1210/jc.2007-1876. Epub 2007 Dec 26. PMID 18160467
- [Background] Howe TE, Shea B, Dawson LJ, Downie F, Murray A, Ross C, Harbour RT, Caldwell LM, Creed G. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD000333. doi: 10.1002/14651858.CD000333.pub2. PMID 21735380
- [Background] Watson SL, Weeks BK, Weis LJ, Horan SA, Beck BR. Heavy resistance training is safe and improves bone, function, and stature in postmenopausal women with low to very low bone mass: novel early findings from the LIFTMOR trial. Osteoporos Int. 2015 Dec;26(12):2889-94. doi: 10.1007/s00198-015-3263-2. Epub 2015 Aug 5. PMID 26243363
- [Background] Weeks BK, Beck BR. The BPAQ: a bone-specific physical activity assessment instrument. Osteoporos Int. 2008 Nov;19(11):1567-77. doi: 10.1007/s00198-008-0606-2. Epub 2008 Apr 15. PMID 18414964
- [Background] Harlow SD, Gass M, Hall JE, Lobo R, Maki P, Rebar RW, Sherman S, Sluss PM, de Villiers TJ; STRAW + 10 Collaborative Group. Executive summary of the Stages of Reproductive Aging Workshop + 10: addressing the unfinished agenda of staging reproductive aging. J Clin Endocrinol Metab. 2012 Apr;97(4):1159-68. doi: 10.1210/jc.2011-3362. Epub 2012 Feb 16. PMID 22344196
- [Derived] Alexander CJ, Kaluta L, Whitman PW, Billington EO, Burt LA, Gabel L. Strength training for osteoporosis prevention during early menopause (STOP-EM): a pilot study protocol for a single centre randomised waitlisted control trial in Canada. BMJ Open. 2025 Feb 5;15(2):e093711. doi: 10.1136/bmjopen-2024-093711. PMID 39909519